CLINICAL TRIAL: NCT04007705
Title: Effects of an Anti-inflammatory Nutritional Intervention in Disease Assessment Parameters, Inflammatory Markers, and Quality of Life of Patients With Fibromyalgia
Brief Title: Anti-inflammatory Nutritional Intervention in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Portuguese Institute of Rheumatology (Unknown); Centro de Investigação Interdisciplinar Egas Moniz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIDFM2019
Record Dates: First submitted 2019-06-04; First posted 2019-07-05 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Fibromyalgia
Keywords: Antiinflammatory diet; Low FODMAPs diet; Gluten, casein, sugar and processed-foods free diet; Nutrition
MeSH Terms: conditions — Fibromyalgia | interventions — Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory and low FODMAPs diet (Experimental): The anti-inflammatory diet is characterized by the exclusion of potential inflammatory foods, such as gluten, dairy and processed food, for three months. During the first month, a low FODMAPs diet will be implemented, followed by the reintroduction of all fruits and vegetables over a consecutive period of 2 months. Additionally, some potentially anti-inflammatory foods will be promoted: Omega-3 through specific fish (tuna fish, salmon, sardine, horse mackerel) and nuts, antioxidant rich foods, such as fruit and vegetables, and the maintenance of glycemic index.
  Interventions: Behavioral: Anti-inflammatory and low FODMAPs diet
- Control (Active Comparator): Dietary counselling based on general recommendations for healthy eating according to the World Health Organization
  Interventions: Behavioral: General healthy eating

INTERVENTIONS:
Behavioral: Anti-inflammatory and low FODMAPs diet — Exemption of the intake of potentially inflammatory foods, namely gluten, dairy and processed foods, over a consecutive period of 3 months. During the first month, a low FODMAPs diet will be implemented, along with the anti-inflammatory diet, followed by the reintroduction of all fruits and vegetables over a consecutive period of 2 months.
  Arms: Anti-inflammatory and low FODMAPs diet
Behavioral: General healthy eating — Healthy eating counseling according to the World Health Organization
  Arms: Control

SUMMARY:
This is a randomized clinical trial, aimed to analyse the effects of a potentially anti-inflammatory nutritional intervention in disease assessment parameters, inflammatory markers, and quality of life of Fibromyalgia patients. Patients in the intervention group will adopt an anti-inflammatory diet and a diet with a low ingestion of fermentable oligo-, di- and monosaccharides, and polyols (FODMAPs), for a 3 months period. Group control will adopt a diet based on general recommendations for healthy eating in accordance with the World Health Organization.

DETAILED DESCRIPTION:
The presence of low grade intestinal inflammation has been reported in Fibromyalgia (FM) patients. Other studies associate the persistence of symptoms described in FM to possible alterations of the intestinal microbiota composition, i.e. dysbiosis, with consequent existence of Small Intestinal Bacterial Overgrowth (SIBO). A sample of 100 female patients diagnosed with FM, followed-up at Portuguese Rheumathology Institute in Lisbon, will be distributed randomly in two groups. Group 1 will adopt an anti-inflammatory diet, which is characterized by the exemption of the intake of potentially inflammatory foods, namely gluten, dairy and ultra-processed foods, over a consecutive period of 3 months. During the first month, a low FODMAPs diet will be implemented, along with the anti-inflammatory diet, followed by the reintroduction of all fruits and vegetables over a consecutive period of 2 months, for a total of 3 months of intervention. Group 2 will adopt a diet based on general recommendations for healthy eating in accordance with the World Health Organization. The Ethics Committee of the Portuguese Institute of Rheumathology approved this intervention study.

The results of this study are expected to determine whether a change in patient nutrition helps to alleviate symptoms, which would optimize medical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FM performed by the physician, according to the Rome III criteria of the American College of Rheumatology, revised in 2010;
* Ability to read and sign the Informed Consent;
* Stable dose therapy within 4 weeks before study start.

Exclusion Criteria:

* Patients with pathologies that prevent the follow-up of the given dietary protocol;
* Patients currently undergoing lactation or pregnancy;
* Prior or current clinical history of abuse of drug or other substances;
* Change of therapy during the intervention period;
* Presence of other inflammatory diseases;
* Uncontrolled medical conditions (eg. Diabetes Mellitus, decompensated heart disease, renal failure, neoplastic diseases, liver diseases).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Change in pain, accessed by Visual Analogue Pain Scale | 1 and 3 months after baseline
  Accessed by Visual Analogue Pain Scale (1 question about pain intensity over the last month, score: 0-10, with 0 = a total pain relief and 10=the greatest pain ever felt).
Change in pain, accessed by Brief Pain Inventory | 1 and 3 months after baseline
  Accessed by Brief Pain Inventory (12 questions about pain severity and pain interference; presented with 0-10 scales, with 0=no interference and 10=interferes completely; scale range from 0 to 120 - higher range represent a worst result).
Change in quality of life accessed by Revised Fibromyalgia Impact Questionnaire | 1 and 3 months after baseline
  Accessed by Revised Fibromyalgia Impact Questionnaire (20 questions about physical functioning (score 0-3, with 0 = optimal and 3 = worst), and about work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression (score 1-10, with 1 = optimal and 10 = worst; scale range from 0 to 117 - higher range represent a worst result).
Change in quality of life accessed by Short-form 36 | 1 and 3 months after baseline
  Accessed by Short-form 36 (36 questions related to the last month, distributed in 8 dimensions: physical function (Score 1-3, with 1 = very limited and 3 = not limited), physical performance, pain, general health, vitality, social function, emotional performance and mental health (score 1-5, with 1 = bad and 5-optimal); scale range from 36 to 142 - higher range represent a worst result).
Change in inflammatory parameters accessed by serum C-reactive protein measurement | 3 months after baseline
  Measurement of serum C-reactive protein (mg/L).
Change in inflammatory parameters accessed by serum erythrocyte sedimentation rate measurement | 3 months after baseline
  Measurement of serum erythrocyte sedimentation rate (mm/h).
Change in inflammatory parameters accessed by serum interleukin-8 measurement | 3 months after baseline
  Measurement of serum and interleukin-8 (pg/mL).

SECONDARY OUTCOMES:
Change in fatigue accessed by Fatigue Severity Survey | 1 and 3 months after baseline
  Accessed by 1 questionnaire: Fatigue Severity Survey (7 questions with scale from 1 to 7, with 1 = fully disagree and 7 = fully agree; scale range from 7 to 49 - higher range represent a worst result).
Change in gastrointestinal symptoms accessed by Visual Analog Scale from a list of common gastrointestinal symptoms | 1 and 3 months after baseline
  Accessed by questionnaire: Visual Analog Scale from a list of common gastrointestinal symptoms (10 questions about gastrointestinal discomfort over the last month, score: 0-10, with 0 = none and 10 = a big discomfort; scale range from 0 to 100 - higher range represent a worst result).
Change in quality of sleep accessed by Pittsburgh Sleep Quality Index | 1 and 3 months after baseline
  Accessed by 1 questionnaire: Pittsburgh Sleep Quality Index (18 questions with a scale from 1 to 4, with 1=no sleep disturbance and 4=to much sleep disturbance; scale range from 18 to 72 - higher range represent a worst result).
Change in weight | 3 months after baseline
  Measurement of weight in Kilograms.
Change in waist circumference | 3 months after baseline
  Measurement of waist circumference in centimeters.
Change in body fat mass | 3 months after baseline
  Measurement by bio-impedance of body fat mass in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rita Silva, MD, Principal Investigator — Universidade do Porto
Locations (1):
- Instituto Português de Reumatologia, Lisbon, Portugal

REFERENCES:
- [Result] Uceyler N, Hauser W, Sommer C. Systematic review with meta-analysis: cytokines in fibromyalgia syndrome. BMC Musculoskelet Disord. 2011 Oct 28;12:245. doi: 10.1186/1471-2474-12-245. PMID 22034969
- [Result] Silva AR, Bernardo A, Costa J, Cardoso A, Santos P, de Mesquita MF, Vaz Patto J, Moreira P, Silva ML, Padrao P. Dietary interventions in fibromyalgia: a systematic review. Ann Med. 2019;51(sup1):2-14. doi: 10.1080/07853890.2018.1564360. PMID 30735059
- [Result] Statovci D, Aguilera M, MacSharry J, Melgar S. The Impact of Western Diet and Nutrients on the Microbiota and Immune Response at Mucosal Interfaces. Front Immunol. 2017 Jul 28;8:838. doi: 10.3389/fimmu.2017.00838. eCollection 2017. PMID 28804483
- [Result] Shivappa N, Steck SE, Hurley TG, Hussey JR, Hebert JR. Designing and developing a literature-derived, population-based dietary inflammatory index. Public Health Nutr. 2014 Aug;17(8):1689-96. doi: 10.1017/S1368980013002115. Epub 2013 Aug 14. PMID 23941862
- [Derived] Silva AR, Bernardo A, de Mesquita MF, Vaz-Patto J, Moreira P, Silva ML, Padrao P. An anti-inflammatory and low fermentable oligo, di, and monosaccharides and polyols diet improved patient reported outcomes in fibromyalgia: A randomized controlled trial. Front Nutr. 2022 Aug 15;9:856216. doi: 10.3389/fnut.2022.856216. eCollection 2022. PMID 36091254
- [Derived] Silva AR, Bernardo A, de Mesquita MF, Vaz Patto J, Moreira P, Silva ML, Padrao P. A study protocol for a randomized controlled trial of an anti-inflammatory nutritional intervention in patients with fibromyalgia. Trials. 2021 Mar 9;22(1):198. doi: 10.1186/s13063-021-05146-3. PMID 33743794